CLINICAL TRIAL: NCT06486688
Title: Virtual SBIRT for Pediatric Primary Care: Increasing Access to Screening, Brief Intervention and Referral to Treatment for Alcohol and Other Drug Use Via Telehealth
Brief Title: Centralized Virtual SBIRT for Pediatric Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1951166
Record Dates: First submitted 2024-06-19; First posted 2024-07-03 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Adolescent Alcohol Use; Mental Health Issue; Alcohol Related Disorders; Adolescents
Keywords: Adolescents; Alcohol; SBIRT; Screening; Drug
MeSH Terms: conditions — Underage Drinking; Alcohol-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care/Traditional SBIRT (Active Comparator): Clinics where appointment-based brief interventions are delivered by a behavioral health clinician assigned to the clinic (Traditional SBIRT arm)
  Interventions: Behavioral: Centralized Virtual SBIRT
- CV SBIRT (Experimental): Clinics where brief interventions are delivered virtually by video or telephone by a centralized behavioral health clinician (CV-SBIRT arm)
  Interventions: Behavioral: Centralized Virtual SBIRT

INTERVENTIONS:
Behavioral: Centralized Virtual SBIRT — Brief interventions are delivered virtually by video or telephone by a centralized behavioral health clinician

SUMMARY:
Adolescent alcohol and other drug (AOD) use is a significant public health problem which contributes to high levels of mortality, morbidity and healthcare costs in young people, and identification and early intervention for these problems is critical to improving outcomes. Screening, Brief Intervention and Referral to Treatment (SBIRT) in pediatric primary care is an evidence-based strategy for addressing these problems, but has not been widely and systematically implemented, for a variety of reasons, including lack of training and staffing resources to support its implementation. This pragmatic, Type 1 Hybrid Comparative Effectiveness Implementation study will examine whether a centralized, virtually-delivered modality of SBIRT, rapidly accessible by multiple pediatric primary care clinics, can be cost-effectively implemented to improve early identification and treatment for AOD use and comorbid mental health problems among adolescents identified as being at high or severe risk of AOD use disorder during adolescent Well Visits.

DETAILED DESCRIPTION:
Adolescent alcohol and other drug (AOD) use is a major public health concern posing significant challenges to healthcare providers, patients and families. It is associated with comorbid psychiatric and medical conditions, poor educational and employment outcomes, accidents and injuries, and avoidable health services utilization and costs (e.g., emergency and inpatient). Early AOD use initiation is associated with alcohol use disorders in adulthood. Screening, Brief Intervention and Referral to Treatment (SBIRT) delivered in pediatric primary care is an effective approach to early identification and intervention and can reduce both AOD use and consequences and co-occurring mental health symptoms, yet widespread implementation is lacking, due to a variety of barriers, including the time constraints and competing priorities faced by pediatricians and lack of trained staff. Research on efficient and cost-effective modalities of SBIRT delivery in pediatric primary care is critical to expanding the evidence base and supporting broader implementation. Accelerated by the pandemic, behavioral telemedicine approaches to addressing adolescent AOD use, and mental health problems are gaining momentum and offer the potential to increase the reach and impact of SBIRT in pediatric primary care. This study's objective is to examine whether a centralized, virtually delivered modality of SBIRT, rapidly accessible by multiple pediatric primary care clinics, can be cost-effectively implemented to improve early identification and treatment for AOD and comorbid mental health problems among adolescents at high or severe risk of AOD use disorder. In this wholly pragmatic, Type 1 Hybrid Comparative Effectiveness Implementation study, set in a large, real-world health system with a highly diverse population, we will compare outcomes in two models of busy, general pediatric primary care clinics with an eligible population of approximately 22,320 12-17 year old adolescents: 1) clinics where brief interventions are delivered virtually by video or telephone by a centralized behavioral health clinician (CV-SBIRT arm), or 2) clinics where appointment-based brief interventions are delivered by a behavioral health clinician assigned to the clinic (Traditional SBIRT arm).

ELIGIBILITY:
Inclusion Criteria:

• The sample will include all adolescents aged 12 through 17 years seen for a Well Visit, who are at risk of AOD use disorder defined as endorsing monthly or more frequent AOD use OR any AOD use and past-two-week depressive symptoms or suicidality.

Exclusion Criteria:

• N/A - all adolescents with a Well Visit are eligible

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22320 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Referrals to behavioral health clinicians for SBIRT | During the 2 year intervention period
  Patients seen by behavioral health clinicians in both intervention arms will be determined via appointment codes
Brief Interventions | During the 2-year intervention period
  Brief Interventions will be documented in the Electronic Health Record via administrative Z-codes within 1 week of the index screening visit.
Referrals | During the 2-year intervention period
  Referrals to specialty treatment will be coded using the electronic referral program in the Electronic Health Records within 1 week of the Brief Intervention.
Specialty Treatment Initiation | Within 2 months of the index screening visit.
  Initiation is defined as at least 1 visit to specialty treatment (Addiction Medicine or Child & Adolescent Psychiatry).
Specialty Treatment Engagement | Within 34 days of the initial specialty care initiation encounter.
  Engagement is defined as 2 or more specialty treatment encounters.
AOD and Mental Health Diagnoses | within 1 year and 2 years of the index screening visit
  Clinical International Classification of Diseases-10 AOD, depression, and anxiety diagnoses
Alcohol and other drug use | 1- and 2-year follow-up visits.
  Alcohol and other drug use will be measured by the Screening to Brief Intervention (S2BI) screening tool: "In the past year, how many times have you used: alcohol, marijuana (smoked, edible, dabs), tobacco (cigarettes), vaping nicotine, vaping marijuana, other substances?" Responses: never, once or twice, monthly, weekly or more
Depressive symptoms | 1- and 2-year follow-up visits.
  Prior two-week depression measures via the Patient Health Questionnaire-2, a validated and commonly used screener for depression: "Over the last 2 weeks how often have you been bothered by the following problems? 1)Little interest or pleasure in doing things; 2) Feeling down, depressed or hopeless?" - Responses: not at all, several days, more than half the days, nearly every day
Suicidality | 1- and 2-year follow-up visits.
  Suicidality measured by: Have you thought seriously about killing yourself, made a plan, or tried to kill yourself? Responses: Y/N
Health Services Utilization | Within 1 year and 2 years of the index screening visit.
  The number of inpatient and Emergency Department encounters

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Division of Research, Pleasanton, California, United States

IPD SHARING:
Plan to Share IPD: No